CLINICAL TRIAL: NCT05044754
Title: Salvage Cryoablation of the Prostate (SCAP) vs High Intensity Focal Ultrasounds (HIFU) for Recurrent Prostate Cancer After Radiation Therapy
Brief Title: SCAP vs HIFU for Recurrent Prostate Cancer After Radiation Therapy
Acronym: SALVPROST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Virgen de las Nieves (Other)
Collaborators: Hospital Universitario Reina Sofia de Cordoba (Other Government); Hospitales Universitarios Virgen del Rocío (Other); Institut Universitaire du Cancer de Toulouse (Other)
Responsible Party: Principal Investigator, Ignacio Puche Sanz, MD PhD Urologist, University Hospital Virgen de las Nieves
Other Study IDs: SALVPROST-YAU-21
Record Dates: First submitted 2021-09-01; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Cryotherapy; High Intensity Focused Ultrasounds; Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — SREBP cleavage-activating protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SCAP: Patients with recurrent prostate cancer undergoing SCAP
  Interventions: Procedure: Local treatment of the prostate (SCAP or HIFU)
- HIFU: Patients with recurrent prostate cancer undergoing HIFU
  Interventions: Procedure: Local treatment of the prostate (SCAP or HIFU)

INTERVENTIONS:
Procedure: Local treatment of the prostate (SCAP or HIFU) — Once the local involvement of the recurrent prostate cancer is confirmed, patient will undergo local treatment of the prostate (SCAP or HIFU)

SUMMARY:
The evidence base relating to the use of SCAP and HIFU is poor, with significant uncertainties relating to long-term oncological outcomes. One of the main limitations when the few studies reported are analyzed is the lack of information about the histopathology both before starting treatment and at the time of recurrence after cryotherapy. The vast majority of studies refer only to BCR-free survival as end point, thus limiting interpretation of real oncological performance of this technique. Furthermore, side effects vary widely from study to study and there are uncertainties about the real morbidity associated to cryotherapy in the salvage setting.

Another important hot issue in this scenario is the potential benefit that new imaging and diagnosis techniques (MRI, targeted biopsy, PSMA) may add for a more accurate indication. This could provide the possibility of better results for SCAP. The clinical value of this new diagnostic tools is unknown in this scenario and needs to be explored.

ELIGIBILITY:
Inclusion Criteria:

* Patients with local recurrence (with histological confirmation) after treatment with radiotherapy or brachytherapy without evidence of distant involvement evaluated preferably with PET/PSMA (if not available then Fluciclovine PET/CT or choline PET/CT must be performed).
* Life expectancy >10 years
* Prostate volume < 100cc
* PSA<10 ng/mL
* mpMRI + fusion/systematic biopsy (template suppl 1) o mpMRI ≤cT3a without affecting the bladder neck or the membranous urethra so that the continence mechanisms of the sphincter are not compromised.

Exclusion Criteria:

* Patients with clinically confirmed distant metastasis
* Any previous major rectal surgery
* Clinically significant lower urinary tract or rectal anomalies
* Existing urethral, rectal, or bladder fistulae

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering local recurrence of prostate cancer after primary treatment with radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
DFS-histology | 1 year
  Disease free survival (confirmed by follow-up biopsy)
DFS-image | 1 year
  Disease free survival (confirmed by follow-up PET-CT )
ADT-FS | 5 years
  Androgen deprivation therapy free survival.

SECONDARY OUTCOMES:
BCR free survival | 5 years
  Time free of biochemical recurrence (PSA)
MFS-PET | 5 years f-u
  Metastasis free survival. rate of patients without any metastasis detected on PET-CT.
Complications rate | 1 year
  Rate of early and long-term complications
Continence | 1 year
  Change in continence scores (ICIQ-SF q)
Sexual function | 1 year
  Changes in sexual function (IIEF questionanaire)
Low urinary tract function | 1 year
  Changes in IPSS questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Puche-Sanz, MD, PhD, Principal Investigator — University Hospital Virgen de las Nieves; Enrique Gomez-Gomez, MD, Principal Investigator — Hospital Universitario Reina Sofia de Cordoba
Locations (4):
- Institut Universitaire du Cancer, Toulouse, France
- Spain (3):
  - Hospital Universitario Reina Sofía, Córdoba, Andalusia
  - Hospital Universitario Virgen de las Nieves, Granada, Andalusia
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Undecided